CLINICAL TRIAL: NCT03280186
Title: Measurement of Bladder Function Change In Patients With Spinal Vascular Malformations Before and After Surgical Intervention
Brief Title: Measurement of Bladder Function Change In Patients With SVMs Before and After Surgical Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, ou tongwen, Director of Urology, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: otw-20170908
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Spinal Vascular Disorder Nos; Neurogenic Bladder Dysfunction Nos
Keywords: Spinal Vascular Malformations; Bladder; Surgical intervention; Urodynamics
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients With SVMs (Experimental): Patients with SVMs will be included in the group and undergo surgery.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — The minimally invasive surgical treatment methods and new techniques will be adopted such as spinal superselective angiography, preoperative embolization, intraoperative electrophysiological monitoring, intraoperative angiography, etc.

SUMMARY:
The investigators goal is to create a better understanding of patient with SVMs reported outcomes for bladder management strategies before and after surgery.

DETAILED DESCRIPTION:
Spinal Vascular malformations (SVMs) are complex neurosurgical lesions and account for 3%-4% of all intradural spinal cord mass lesions, which can influence the function of bladder. However, no study show the relationship of the SVMs and bladder function. The investigators goal is to create a better understanding of patient reported outcomes for bladder management strategies before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

- patient diagnosed with spinal vascular diseases including intradural arteriovenous malformation, intradural arteriovenous fistula, dural arteriovenous fistula, extradural arteriovenous malformation, paravertebral arteriovenous malformation, paravertebral arteriovenous fistula, cobbs' syndrome, other spinal arteriovenous metameric syndromes involve the spinal cord. patient not received surgical or interventional treatment before patient with normal cardiac, renal and hepatic function patient capable of understanding the content of the patient information / Informed Consent Form patient willing and able to participate in the registry

Exclusion Criteria:

- patient received surgical treatment or interventional treatment before patient is pregnant patient allergic to iodine patient unable to complete follow-up patient with cerebral lesions patient with other spinal lesions patient with cardiac, renal or hepatic dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
bladder function change in urodynamics | postoperative 3 months and 12 months
  bladder function will be better in urodynamics after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Tongwen Ou, M.D, Study Director — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No